CLINICAL TRIAL: NCT02337036
Title: Building a Population Pharmacokinetic Model of Tacrolimus in Paediatric Liver Transplant Patients
Brief Title: Pharmacokinetic of Tacrolimus in Paediatric Liver Transplant Patients
Acronym: TACTHEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P120904; 2013-000948-26 (EudraCT Number)
Record Dates: First submitted 2014-12-05; First posted 2015-01-13 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Liver Transplantation, Child
Keywords: Liver transplantation; Child; Tacrolimus; Pharmacokinetic
MeSH Terms: interventions — Pharmacogenomic Variants; Pharmacogenomic Testing; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: Pharmacokinetic and Pharmacogenetic (Experimental): Liver Transplant Children treated with tacrolimus
  Interventions: Other: Pharmacokinetic; Other: Pharmacogenetic; Drug: Tacrolimus

INTERVENTIONS:
Other: Pharmacokinetic — Taking blood samples for an Pharmacokinetic of tacrolimus in Paediatric Liver Transplant Patients treated with tacrolimus
Other: Pharmacogenetic — Pharmacogenetic study
Drug: Tacrolimus — These Patients are treated with tacrolimus after the Liver Transplantation

SUMMARY:
Tacrolimus is the cornerstone immunosuppressant in children with liver transplantation, its use is complicated by its narrow therapeutic index and variable pharmacokinetics. This study is designed to assess the posology of tacrolimus in post-transplantation in the month after liver transplantation to obtain a therapeutic target between 10-15 ng/mL and the impact of biological and genetic factors on the pharmacokinetic parameters in paediatric liver transplant recipients.

DETAILED DESCRIPTION:
Tacrolimus is the cornerstone immunosuppressant in children with liver transplantation, its use is complicated by its narrow therapeutic index and variable pharmacokinetics. Therapeutic drug monitoring (TDM) of tacrolimus, based on whole-blood trough concentration (C0) values, is mandatory for use of twice-daily tacrolimus (Prograf_) as in order to decrease interindividual variability in exposure and thereby minimize the risk of acute rejection and the occurrence of adverse effects (mainly nephrotoxicity and, to a lesser extent, neurotoxicity).

Until now, the C0 is the easiest means of individual dose adjustment, as only one blood sample is required and the clinician can easily calculate the dose needed to reach the target. Many factors have an impact on the pharmacokinetic parameters. However the adaptation of the time to achieve the target stays an issue. Among factors of inter and intra variability of pharmacokinetic of tacrolimus, some of them are specific of the pediatric liver transplantation population.

Aims: To build a population pharmacokinetic model that describes the apparent clearance of tacrolimus and the potential demographic, clinical and genetically controlled factors that could lead to inter-patient pharmacokinetic variability within children following liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age of children who need to have a liver transplantation : between 6 month and 12 years
* Formulary of consent signed by the two parents.
* Children who need to receive tacrolimus per os (Modigraf® ) only after liver transplantation associated to Simulect® (basilixumab) in post-transplantation immediately as main
* Affiliation to the system of social protection.

Exclusion Criteria:

* Children who need a multi organs transplantation
* Hypersensibility or Contraindication to Modigraf® or others macrolides.
* Patients retransplanted in the 14 days after the transplantation
* Patients with multivisceral failure
* Patients who have an introduction of tacrolimus 3 days after transplantation
* Patients who need complementary immunosuppressive drugs with corticoids excepted methylprednisolone used for reject
* Patients who received Prograf® per os or iv.
* Patients who received Cellcept® or Myfortic®
* Opposition to sign the formulary of consent or the understand the note of information

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2013-12; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Blood concentration of tacrolimus (ng/mL) | Between day2 and day4 and day 10 and day14, after day 21
  Residual concentration, Cmin, Cmax, Cl/F and Area Under the Curve of tacrolimus (AUC)

SECONDARY OUTCOMES:
"P3A5" cytochrome (CYP3A5/4), "ABCB1" genotypes of donor and recipient. | Up to 3 years
Factor V and prothrombin time | Up to 3 years
  To estimate a delayed graft function
Time to achieve two concentrations of tacrolimus in the therapeutic target without change of posology | Up to 3 years
Clinical Occurrence of adverse events (reject and/or adverse effects with tacrolimus) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel GONZALES, PhD, MD, Principal Investigator — AP-HP, Bicêtre Hospital
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France